CLINICAL TRIAL: NCT01046890
Title: Drug Interactions Between Echinacea Purpurea and Darunavir/Ritonavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: IrsiCaixa (Other); Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQUIDAR
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Darunavir; Echinacea purpurea; Interaction; Complementary Therapies
MeSH Terms: conditions — HIV Infections | interventions — Echinacea extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- darunavir/ritonavir + root of Echinacea purpurea (Experimental): darunavir/ritonavir + root of Echinacea purpurea
  Interventions: Drug: Echinacea

INTERVENTIONS:
Drug: Echinacea — darunavir/ritonavir 600/100 mg + root of Echinacea purpurea 500 mg every 6 hours
  Other Names: N/H

SUMMARY:
The purpose of this clinical trial is to characterize drug interactions between one medicinal herb widely used by HIV infected patients: Echinacea sp. and the protease inhibitor darunavir/ritonavir.

DETAILED DESCRIPTION:
15 patients on antiretroviral therapy with darunavir/ritonavir 600/100 mg twice a day during four weeks will be recruited. The patients will receive treatment with Echinacea purpurea for 14 days, 500 mg every 6 hours. A 12 hour pharmacokinetic curve will be obtained at baseline and on day 14.

ELIGIBILITY:
Inclusion Criteria:

1. Patients infected with HIV-1 (at least one documented positive Western-Blot).
2. Age =/+ 18 years.
3. Patients receiving antiretroviral therapy containing darunavir / ritonavir at the approved dose of 600/100 mg twice daily for at least 4 weeks
4. HIV viral load in plasma <50 copies / mL
5. Absence of acute infections and / or tumors in the three months prior to inclusion.
6. Subject able to follow the treatment period, without suspicion of poor adherence in previous antiretroviral treatments.
7. Voluntary written informed consent.

Exclusion Criteria:

1. Any clinical or historical observation that could interfere with the pharmacokinetics of medications, such as gastrointestinal illness or surgery (except for herniotomy and appendectomy), changes in the composition of plasma proteins, some indication of hepatic or renal dysfunction.
2. Active alcohol consumption (> 50 g / day) or illicit drugs (except cannabis).
3. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
plasma concentration of darunavir and ritonavir | DAY 14

SECONDARY OUTCOMES:
Clearance (CL/F) | DAY 14
Volume of distribution (V/F) | DAY 14
Elimination half-life (t1/2) | DAY 14
Area under the plasma concentration-time curve during the dosing interval | DAY 14
Adverse events and laboratory alterations | DAY 14
HIV Viral load in plasma | DAY 14

CONTACTS AND LOCATIONS:
Overall Officials: Jose Moltó, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation, HIV Unit
Locations (1):
- Lluita contra la Sida Foundation, HIV Unit, Irsi Caixa Foundation, Badalona, Spain